CLINICAL TRIAL: NCT02222714
Title: A Multi-center, Phase 2 Study Using a Continual Reassessment Method to Determine the Safety and Tolerability of 3K3A-APC in Combination With tPA, Mechanical Thrombectomy or Both in Moderate to Severe Acute Ischemic Stroke
Brief Title: Safety Evaluation of 3K3A-APC in Ischemic Stroke
Acronym: RHAPSODY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ZZ Biotech, LLC (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Cedars-Sinai Medical Center (Other); Massachusetts General Hospital (Other); University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZZ-3K3A-201 (NN104); 1U01NS088312-01 (NIH); U01NS077352 (NIH); U01NS077179-01 (NIH)
Record Dates: First submitted 2014-08-18; First posted 2014-08-21 (Estimated); Results first posted 2018-11-08 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-10

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; stroke; APC; 3K3A; 3K3A-APC; activated protein C; RHAPSODY
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — 3K3A-APC protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 120 µg/kg of 3K3A-APC (Active Comparator): 3K3A-APC, q12h for up to 5 doses
  Interventions: Biological: 3K3A-APC
- 240 µg/kg of 3K3A-APC (Active Comparator): 3K3A-APC, q12h for up to 5 doses
  Interventions: Biological: 3K3A-APC
- 360 µg/kg of 3K3A-APC (Active Comparator): 3K3A-APC, q12h for up to 5 doses
  Interventions: Biological: 3K3A-APC
- 540 µg/kg of 3K3A-APC (Active Comparator): 3K3A-APC, q12h for up to 5 doses
  Interventions: Biological: 3K3A-APC
- Placebo (Placebo Comparator): Matching placebo, q12h for up to 5 doses
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: 3K3A-APC — 3K3A-APC, diluted in 0.9% sodium chloride in water, given as 100 mL IV infusion
  Other Names: 3K3A-Activated Protein C
  Arms: 120 µg/kg of 3K3A-APC; 240 µg/kg of 3K3A-APC; 360 µg/kg of 3K3A-APC; 540 µg/kg of 3K3A-APC
Drug: Placebo — Matching placebo, 0.9% sodium chloride in water, given as 100 mL IV infusion
  Other Names: Matching Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the safety, pharmacokinetics (PK) and preliminary efficacy of multiple ascending intravenous doses of 3K3A-APC, a Recombinant Variant of Human activated protein C (APC), in in the treatment of acute ischemic stroke following treatment with recombinant tissue plasminogen activator (tPA), mechanical thrombectomy or both.

DETAILED DESCRIPTION:
This was a multicenter, prospective, randomized, controlled, double-blinded Phase 2 study intended to evaluate the safety, PK and preliminary efficacy of 3K3A-APC following treatment with tPA, mechanical thrombectomy or both in subjects with moderate to severe acute ischemic stroke.

Approximately 115 subjects were to be randomized, which included the planned 88 subjects in groups of 4 subjects to either 3K3A-APC or placebo (in a 3:1 ratio) and the additional placebo subjects who were enrolled during safety review pauses. This study used a modified version of the continual reassessment method (CRM) in order to establish a maximum tolerated dose (MTD).

Eligible subjects received 3K3A-APC or placebo every 12 hours for up to 5 doses (approximately 3 days), or until discharge from the hospital, whichever occurred first. Subjects were monitored for safety evaluations through Day 7 (or discharge, if earlier) and were expected to be seen on Day 7, 14, 30, and 90 for safety and outcome evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke
* Able to receive IV tPA, mechanical thrombectomy or both
* National Institutes of Health Stroke Scale (NIHSS) score of ≥ 5
* Signed informed consent
* Mechanical thrombectomy subjects only: onset time to arterial puncture time < 6 hours

Exclusion Criteria:

* History of stroke or penetrating head injury within 90 days prior to enrollment
* History of previous or current diagnosis of intracranial hemorrhage that represents a potential for re-hemorrhage if subjected to thrombolytic therapy or mechanical thrombectomy
* Moyamoya disease, cerebral arterio-venous malformation (AVM), known unsecured aneurysm requiring intervention during the acute study period
* Presence of other neurological or non-neurological co-morbidities that may lead, independently of the current stroke, to further deterioration in the subject's neurological status during the trial period
* Presence of premorbid neurological deficits and functional limitations assessed by a retrospective Modified Rankin Scale (mRS) score of ≥ 2
* Mechanical thrombectomy subjects only: baseline non-contrast CT scan revealing a large core occlusion as defined by local protocol
* Prolonged prothrombin time (PT) or activated partial thromboplastin time (aPTT)
* Severe hypertension or hypotension
* Glomerular filtration rate (GFR) <35 mL/min
* Blood glucose concentration < 50 mg/dL
* Prior exposure to any exogenous form of APC

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-10; Primary Completion 2017-04-18 (Actual); Study Completion 2017-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick D. Lyden, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (15):
- United States (15):
  - Stroke Center, Los Angeles, California
  - Stroke Center, Chicago, Illinois
  - Stroke Center, Kansas City, Kansas
  - Stroke Center, Boston, Massachusetts
  - Stroke Center, St Louis, Missouri
  - Stroke Center, Buffalo, New York
  - Stroke Center, New York, New York
  - Stroke Center, Rochester, New York
  - Stroke Center, Cincinnati, Ohio
  - Stroke Center, Columbus, Ohio
  - Stroke Center, Pittsburgh, Pennsylvania
  - Stroke Center, Nashville, Tennessee
  - Stroke Center, Dallas, Texas
  - Stroke Center, Salt Lake City, Utah
  - Stroke Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lyden P, Levy H, Weymer S, Pryor K, Kramer W, Griffin JH, Davis TP, Zlokovic B. Phase 1 safety, tolerability and pharmacokinetics of 3K3A-APC in healthy adult volunteers. Curr Pharm Des. 2013;19(42):7479-85. doi: 10.2174/1381612819666131230131454. PMID 24372304
- [Derived] Lyden P, Pryor KE, Coffey CS, Cudkowicz M, Conwit R, Jadhav A, Sawyer RN Jr, Claassen J, Adeoye O, Song S, Hannon P, Rost NS, Hinduja A, Torbey M, Lee JM, Benesch C, Rippee M, Rymer M, Froehler MT, Clarke Haley E, Johnson M, Yankey J, Magee K, Qidwai J, Levy H, Mark Haacke E, Fawaz M, Davis TP, Toga AW, Griffin JH, Zlokovic BV; NeuroNEXT Clinical Trials Network NN104 Investigators. Final Results of the RHAPSODY Trial: A Multi-Center, Phase 2 Trial Using a Continual Reassessment Method to Determine the Safety and Tolerability of 3K3A-APC, A Recombinant Variant of Human Activated Protein C, in Combination with Tissue Plasminogen Activator, Mechanical Thrombectomy or both in Moderate to Severe Acute Ischemic Stroke. Ann Neurol. 2019 Jan;85(1):125-136. doi: 10.1002/ana.25383. Epub 2019 Jan 7. PMID 30450637
- [Derived] Lyden P, Weymer S, Coffey C, Cudkowicz M, Berg S, O'Brien S, Fisher M, Haley EC, Khatri P, Saver J, Levine S, Levy H, Rymer M, Wechsler L, Jadhav A, McNeil E, Waddy S, Pryor K. Selecting Patients for Intra-Arterial Therapy in the Context of a Clinical Trial for Neuroprotection. Stroke. 2016 Dec;47(12):2979-2985. doi: 10.1161/STROKEAHA.116.013881. Epub 2016 Nov 1. PMID 27803392

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 120 µg/kg of 3K3A-APC | 240 µg/kg of 3K3A-APC | 360 µg/kg of 3K3A-APC | 540 µg/kg of 3K3A-APC | Placebo
Started | 15 | 24 | 12 | 15 | 44
Completed | 15 | 22 | 8 | 11 | 37
Not Completed | 0 | 2 | 4 | 4 | 7
Not completed — Death | 0 | 2 | 3 | 4 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- 120 µg/kg of 3K3A-APC; 240 µg/kg of 3K3A-APC; 360 µg/kg of 3K3A-APC; 540 µg/kg of 3K3A-APC: 3K3A-APC, q12h for up to 5 doses 3K3A-APC: 3K3A-APC, diluted in 0.9% sodium chloride in water, given as 100 mL IV infusion
- Placebo: Matching placebo, q12h for up to 5 doses Placebo: Matching placebo, 0.9% sodium chloride in water, given as 100 mL IV infusion
- Total: Total of all reporting groups
Arm/Group | 120 µg/kg of 3K3A-APC | 240 µg/kg of 3K3A-APC | 360 µg/kg of 3K3A-APC | 540 µg/kg of 3K3A-APC | Placebo | Total
Number analyzed (Participants) | 15 | 24 | 12 | 15 | 44 | 110
Age, Continuous [Mean (Full Range); unit: years] | 63.3 [28 to 84] | 61.4 [33 to 88] | 65.3 [43 to 89] | 66.2 [42 to 89] | 63.8 [44 to 83] | 63.7 [28 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 6 | 8 | 20 | 57
  Male | 4 | 12 | 6 | 7 | 24 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 1 | 7 | 11
  Not Hispanic or Latino | 11 | 22 | 12 | 13 | 36 | 94
  Unknown or Not Reported | 2 | 1 | 0 | 1 | 1 | 5
History of Hypertension [Count of Participants; unit: Participants] | 11 | 21 | 9 | 11 | 33 | 85
History of Diabetes [Count of Participants; unit: Participants] | 6 | 6 | 2 | 4 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events That Meet Dose-limiting Toxicity (DLT) Criteria Specified in Protocol
Description: Specific AEs in the study were defined in the protocol to be dose-limiting toxicity events. Any given patient was adjudicated in a binary way to either have had a DLT or not to have had a DLT.
Time Frame: 48-hours following last dose
Population: Evaluable participants
Measure: Count of Participants; unit: Participants
Arm/Group | 120 µg/kg of 3K3A-APC | 240 µg/kg of 3K3A-APC | 360 µg/kg of 3K3A-APC | 540 µg/kg of 3K3A-APC | Placebo
Number analyzed (Participants) | 15 | 24 | 12 | 15 | 44
Participants
  1-hour post dose aPTT out of range | 0 | 1 | 0 | 0 | 1
  SICH associated with neuroworsening | 0 | 1 | 0 | 0 | 0
  ALT/AST, TBL, ALP, AT values out of range | 0 | 0 | 0 | 0 | 0
  Serious bleeding | 0 | 0 | 0 | 0 | 0
  Abnormal lab value related to study treatment | 0 | 0 | 1 | 0 | 2
  Any other AE leading to cessation of dosing | 0 | 0 | 0 | 0 | 1
  Total | 0 | 2 | 1 | 0 | 4

2. Secondary Outcome: Number of Participants With a Presence of Measurable Bleeds in the Brain (Hemorrhage and Microbleeds) as Determined by 1.5T MRI
Description: MRI examination to include-at minimum-T1 and T2 weighted images, as well as diffusion weighted imaging (DWI) and susceptibility weighted imaging (SWI) sequences. Post-tPA microbleeds-defined as hypointensities less than 5mm in diameter seen on SWI-will be counted as tPA-related only if found within the ischemic territory. All other areas of hypointensity on SWI larger than 5mm diameter will be counted as tPA-related regardless of the territory in which they are found. All treated subjects (regardless of dose) will be compared to all placebo subjects using a Pearson chi-square test.
Time Frame: Day 30
Population: Subjects with a Day 30 scan collected.
Measure: Count of Participants; unit: Participants
Groups:
- 3K3A-APC Total: All 3K3A-APC treated groups combined
- Placebo: Placebo group
Arm/Group | 3K3A-APC Total | Placebo
Number analyzed (Participants) | 43 | 37
Participants
  Hemorrhage (>0.06mL) | 24 | 25
  Microbleed (>0) | 7 | 8

3. Secondary Outcome: PK of 3K3A-APC by Compartmental Analysis (Clearance)
Description: Measured following a single dose; primary parameters (CL, V) were used to fit the model. Secondary parameters (Cmax, AUC(inf), λz, t1/2) were estimated from the primary parameters.
Time Frame: Following a single dose, on Day 1, 2 or 3: End of infusion (EOI) and 20, 40, 60 and 80 minutes following EOI
Population: The PK population included all subjects who had sufficient data for PK analysis, and who had not been excluded from analysis for protocol deviations that could impact the calculation or interpretation of the PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hr
Arm/Group | 120 µg/kg of 3K3A-APC | 240 µg/kg of 3K3A-APC | 360 µg/kg of 3K3A-APC | 540 µg/kg of 3K3A-APC
Number analyzed (Participants) | 5 | 3 | 5 | 8
mL/hr | 20994 (57.1) | 17814 (16.7) | 18504 (49.9) | 24403 (70.5)

4. Secondary Outcome: PK of 3K3A-APC by Compartmental Analysis (Volume of Distribution)
Description: as for outcome 3
Time Frame: Following a single dose, on Day 1, 2 or 3: End of infusion (EOI) and 20, 40, 60 and 80 minutes following EOI
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL
Arm/Group | 120 µg/kg of 3K3A-APC | 240 µg/kg of 3K3A-APC | 360 µg/kg of 3K3A-APC | 540 µg/kg of 3K3A-APC
Number analyzed (Participants) | 5 | 3 | 5 | 8
mL | 8242 (46.9) | 6051 (25.6) | 7164 (79.0) | 11437 (125)

5. Secondary Outcome: PK of 3K3A-APC by Compartmental Analysis (Cmax)
Description: as for outcome 3
Time Frame: Following a single dose, on Day 1, 2 or 3: End of infusion (EOI) and 20, 40, 60 and 80 minutes following EOI
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 120 µg/kg of 3K3A-APC | 240 µg/kg of 3K3A-APC | 360 µg/kg of 3K3A-APC | 540 µg/kg of 3K3A-APC
Number analyzed (Participants) | 5 | 3 | 5 | 8
ng/mL | 0.957 (59.1) | 2.37 (11.0) | 2.80 (77.6) | 3.32 (138)

6. Secondary Outcome: PK of 3K3A-APC by Compartmental Analysis (AUC[0-inf])
Description: as for outcome 3
Time Frame: Following a single dose, on Day 1, 2 or 3: End of infusion (EOI) and 20, 40, 60 and 80 minutes following EOI
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr▪ng/mL
Arm/Group | 120 µg/kg of 3K3A-APC | 240 µg/kg of 3K3A-APC | 360 µg/kg of 3K3A-APC | 540 µg/kg of 3K3A-APC
Number analyzed (Participants) | 5 | 3 | 5 | 8
hr▪ng/mL | 0.513 (64.7) | 1.16 (6.79) | 1.49 (56.1) | 2.06 (92.7)

7. Secondary Outcome: PK of 3K3A-APC by Compartmental Analysis (λz)
Description: as for outcome 3
Time Frame: Following a single dose, on Day 1, 2 or 3: End of infusion (EOI) and 20, 40, 60 and 80 minutes following EOI
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hr
Arm/Group | 120 µg/kg of 3K3A-APC | 240 µg/kg of 3K3A-APC | 360 µg/kg of 3K3A-APC | 540 µg/kg of 3K3A-APC
Number analyzed (Participants) | 5 | 3 | 5 | 8
1/hr | 2.55 (13.4) | 2.94 (10.5) | 2.58 (34.9) | 2.13 (45.2)

8. Secondary Outcome: PK of 3K3A-APC by Compartmental Analysis (Half-life)
Description: as for outcome 3
Time Frame: Following a single dose, on Day 1, 2 or 3: End of infusion (EOI) and 20, 40, 60 and 80 minutes following EOI
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | 120 µg/kg of 3K3A-APC | 240 µg/kg of 3K3A-APC | 360 µg/kg of 3K3A-APC | 540 µg/kg of 3K3A-APC
Number analyzed (Participants) | 5 | 3 | 5 | 8
hr | 0.272 (13.4) | 0.235 (10.5) | 0.268 (34.9) | 0.325 (45.2)

ADVERSE EVENTS:
Time Frame: AEs were collected through Study Day 7 and were followed until resolution or a new baseline was established, up to Study Day 90. SAEs were collected through Study Day 30, and were followed until resolution (or resolution with sequelae), up to Study Day 90.
Description: Standard definitions of adverse events and serious adverse events were used.
Arm/Group | 120 µg/kg of 3K3A-APC | 240 µg/kg of 3K3A-APC | 360 µg/kg of 3K3A-APC | 540 µg/kg of 3K3A-APC | 3K3A-APC Total | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 2/24 | 3/12 | 4/15 | 9/66 | 6/44
Serious Adverse Events (participants affected / at risk) | 8/15 | 9/24 | 4/12 | 9/15 | 30/66 | 18/44
Other Adverse Events (participants affected / at risk) | 10/15 | 18/24 | 8/12 | 9/15 | 45/66 | 36/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 120 µg/kg of 3K3A-APC (N=15) | 240 µg/kg of 3K3A-APC (N=24) | 360 µg/kg of 3K3A-APC (N=12) | 540 µg/kg of 3K3A-APC (N=15) | 3K3A-APC Total (N=66) | Placebo (N=44)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 2 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 4 | 0 | 0 | 1 | 5 | 4
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Blood fibrinogen decreased (Investigations) | 0 | 1 | 0 | 2 | 3 | 1
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
Blood sodium increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 1
Troponin increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 1 | 0 | 4 | 5 | 3
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 3 | 0 | 0 | 3 | 2
Cerebrovascular accident (Nervous system disorders) | 1 | 3 | 0 | 1 | 5 | 3
Convulsion (Nervous system disorders) | 2 | 0 | 0 | 0 | 2 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 2 | 0
Aneurysm repair (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 120 µg/kg of 3K3A-APC (N=15) | 240 µg/kg of 3K3A-APC (N=24) | 360 µg/kg of 3K3A-APC (N=12) | 540 µg/kg of 3K3A-APC (N=15) | 3K3A-APC Total (N=66) | Placebo (N=44)
Anaemia (Blood and lymphatic system disorders) | 5 | 4 | 2 | 2 | 13 | 6
Leukocytosis (Blood and lymphatic system disorders) | 0 | 3 | 1 | 2 | 6 | 6
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 5
Constipation (Gastrointestinal disorders) | 0 | 5 | 1 | 0 | 6 | 4
Pyrexia (General disorders) | 1 | 2 | 1 | 0 | 4 | 4
Urinary tract infection (Infections and infestations) | 1 | 5 | 3 | 1 | 10 | 8
Contusion (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0 | 3 | 3
Activated partial thromboplastin time prolonged (Investigations) | 0 | 4 | 0 | 0 | 4 | 2
Blood calcium decreased (Investigations) | 1 | 2 | 1 | 1 | 5 | 1
Blood fibrinogen decreased (Investigations) | 0 | 3 | 0 | 0 | 3 | 4
Lymphocyte count decreased (Investigations) | 2 | 0 | 0 | 1 | 3 | 3
Prothrombin time prolonged (Investigations) | 1 | 3 | 0 | 1 | 5 | 6
Haemorrhage intracranial (Nervous system disorders) | 2 | 4 | 4 | 4 | 14 | 16
Headache (Nervous system disorders) | 1 | 6 | 2 | 3 | 12 | 10
Haematuria (Renal and urinary disorders) | 1 | 0 | 1 | 1 | 3 | 4
Hypotension (Vascular disorders) | 0 | 2 | 1 | 0 | 3 | 3

LIMITATIONS AND CAVEATS:
The study was designed and powered for evaluating DLTs and identifying a maximum tolerated dose, not for efficacy endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-12-07): https://cdn.clinicaltrials.gov/large-docs/14/NCT02222714/SAP_000.pdf
  • Study Protocol (2016-10-07): https://cdn.clinicaltrials.gov/large-docs/14/NCT02222714/Prot_001.pdf